CLINICAL TRIAL: NCT03020862
Title: Beetroot Juice - Effects on Performance in Chronic Obstructive Pulmonary Disease Patients
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D2013A2014
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Obstructive Pulmonary Disease Moderate
Keywords: Dietary nitrate; Physical performance; Blood pressure; Nitrite; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo ---> Dietary beetroot (Experimental): Placebo was administrated in the first period of the cross-over trial, while the intervention beverage Dietary Beetroot juice was administrated in the second period of the trial.
  The placebo: was an NO3- negligble drink from James White Drinks England (Beet-it), which was otherwise similar to the dietary beetroot juice in nutrient composition, smell and appearance. Dose: 2x70 mL consumed twice a day for six days.
  Intervention beverage, Dietary beetroot juice:Consumed as beetroot juice from James White Drinks England (Beet-it) and contained 300 mg dietary nitrate. Dose: 2x70 mL consumed twice a day for six days.
  Interventions: Dietary Supplement: Dietary beetroot juice
- Dietary beetroot juice --> Placebo (Experimental): The intervention beverage Dietary beetroot juice was administrated in the first period of the cross-over trial, while placebo was administrated in the second period of the trail Intervention beverage, Dietary beetroot juice:Consumed as beetroot juice from James White Drinks England (Beet-it) and contained 300 mg dietary nitrate. Dose: 2x70 mL consumed twice a day for six days. The placebo: was an NO3- negligble drink from James White Drinks England (Beet-it), which was otherwise similar to the dietary beetroot juice in nutrient composition, smell and appearance. Dose: 2x70 mL consumed twice a day for six days.
  Interventions: Dietary Supplement: Dietary beetroot juice

INTERVENTIONS:
Dietary Supplement: Dietary beetroot juice — Consumed as concentrated beetroot juice from James White Drinks England (Beet-it) and contained 300 mg dietary nitrate. Dose: 2x70 mL consumed twice a day for six days.

SUMMARY:
The purpose is to evaluate exercise performance in patients with Chronic Obstructive Pulmonary Disease (COPD) after supplementing with higher doses of dietary NO3-, compared to previous studies, as beetroot juice for seven days. The secondary purpose is to evaluate oxygen consumption of submaximal cycling, amendments in blood pressure, and physical activity level.

DETAILED DESCRIPTION:
The purpose is to evaluate exercise performance in patients with Chronic Obstructive Pulmonary Disease (COPD) using the 6-minute walk test (6MWT) after supplementing with higher doses of dietary NO3- compared to previous studies, as beetroot juice for seven days. The secondary purpose is to evaluate oxygen consumption of submaximal cycling, amendments in blood pressure, and physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-severe Chronics Obstructive Pulmonary Disease (COPD) (FEV1 <80% of predicted).

Exclusion Criteria:

* Smoking,
* failure to complete physical testing,
* on-going participation in rehabilitation programs,
* pacemaker or use of nicotine products,
* oxygen mask,
* beta blockers,
* antibacterial mouthwash,
* chewing gum or stomach-neutralizing medicine during the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Physical performance on 6-min walk test (6MWT) | 6 minutes

SECONDARY OUTCOMES:
Blood Pressure | At baseline and 150 minutes after consumption of beverages
Plasma Nitrite concentration | Baseline, 150 and 210 minutes after consumption of beverages
Oxygen consumption during submaximal cycling | Two trials of 6 minutes duration (10 min break between trials)
Physical activity level | Six days
  Measured all intervention days except on the day of testing

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, Principal Investigator — Aarhus University, Department for Public Health, Section for Sport Sciene
Locations (1):
- Sport Science, Department of Public Health, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No